CLINICAL TRIAL: NCT01894776
Title: A Drug Interaction Study Investigating the Effect of Rifabutin on the Pharmacokinetics of Maraviroc
Acronym: RIFAMARA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013 0080-01H
Record Dates: First submitted 2013-06-19; First posted 2013-07-10 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: HIV Infection; HIV-1 Infection; Mycobacterium Avium Complex (MAC)
Keywords: healthy volunteers
MeSH Terms: conditions — HIV Infections; Mycobacterium avium-intracellulare Infection | interventions — Rifabutin; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maraviroc (Experimental): Two period pharmacokinetic drug-drug interaction Period one -Maraviroc alone; Period two -Maraviroc and Rifabutin
  Substance: Maraviroc (Celsentri, MVC) tablets, 300 mg; dose: oral, 300 mg (1 tablet) twice daily
  Substance: Rifabutin (mycobutin, RFB) capsules, 150 mg; dose: oral, 300 mg (2 capsules) once daily
  Interventions: Drug: Rifabutin; Drug: Maraviroc

INTERVENTIONS:
Drug: Rifabutin — Substance: Rifabutin Daily dose: oral, 300 mg once daily (8:00 am) for 10 days
  Other Names: Mycobutin, RFB
Drug: Maraviroc — Substance maraviroc daily dose 300 mg twice daily (8:00 am and 8:00 pm) for 15 days
  Other Names: Celsentri, MVC

SUMMARY:
Healthy volunteers are being recruited for this pharmacokinetics study. The objective is to characterize the pharmacokinetic properties of maraviroc alone and when administered with rifabutin and to assess rifabutin and 25-O-desacetyl-rifabutin pharmacokinetics compared to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign informed consent prior to any study-related activities.
* Male or female participants between 18 and 65 years of age inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Healthy, i.e. not suffering from an acute or chronic illness and not using medications.
* Acceptable medical history, physical examination, and 12-lead ECG at screening.
* Acceptable laboratory values that indicate adequate baseline organ function at screening visit.
* Willing to stop using any herbal or natural health products for 2 weeks prior to and during the study including: Grapefruit, grapefruit juice, St. John's Wort.
* Willingness to abstain from alcohol use for 3 days prior to and during the study.
* Participant must practice a reliable method of birth control while they are participating in the study; for instance an intrauterine device (IUD), condom with spermicidal gel or foam, diaphragm with spermicidal gel or foam, vasectomy, tubal ligation, hysterectomy or abstinence or female must be post menopausal for at least one year.

Exclusion Criteria:

* Have serological evidence of exposure to HIV
* Female patients of childbearing potential who has a positive urine pregnancy test at screening
* Participants not willing to use a reliable method of barrier contraception during the study.
* Is breastfeeding.
* Inability to adhere to protocol.
* Use of any medications (2 weeks prior to or during the study) other than occasional use of acetaminophen.
* Participants taking oral contraceptive medications.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Patients may be excluded from the study for other reasons, at the investigator's discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Cameron, MD, Principal Investigator — The Ottawa Hospital, Ottawa Hospital Research Institute, University of Ottawa
Locations (1):
- The Ottawa Hospital -General Campus, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Ghannad M, Dennehy M, la Porte C, Seguin I, Tardiff D, Mallick R, Sabri E, Zhang G, Kanji S, Cameron DW. A drug interaction study investigating the effect of Rifabutin on the pharmacokinetics of Maraviroc in healthy subjects. PLoS One. 2019 Oct 24;14(10):e0223969. doi: 10.1371/journal.pone.0223969. eCollection 2019. PMID 31647836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Clinical Investigation Unit (CIU) at the OHRI has a database of healthy volunteers interested in participating in clinical studies who were contacted and recruited by phone or email. The first patient was recruited on 06 Sept 2013 and the last follow-up visit was on 23 Dec 2013.
Groups:
- Maraviroc: Two period pharmacokinetic drug-drug interaction Period one -Maraviroc alone; Period two -Maraviroc and Rifabutin
  Substance: Maraviroc (Celsentri, MVC) tablets, 300 mg; dose: oral, 300 mg (1 tablet) twice daily
  Substance: Rifabutin (mycobutin, RFB) capsules, 150 mg; dose: oral, 300 mg (2 capsules) once daily
  Rifabutin: Substance: Rifabutin Daily dose: oral, 300 mg once daily (8:00 am) for 10 days
  Maraviroc: Substance maraviroc daily dose 300 mg twice daily (8:00 am and 8:00 pm) for 15 days
Period: Overall Study
Arm/Group | Maraviroc
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: A single participant dropped out due to Nausea. This resulted in 14 participants Data only being analyzed.
Arm/Group | Maraviroc
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants] — Population: 15 patients underwent baseline measurements and allocated to intervention. However, only 14 were analyzed due to 1 participant withdrawing from the study due to Nausea.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 14
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 15 patients underwent baseline measurements and allocated to intervention. However, only 14 were analyzed due to 1 participant withdrawing from the study due to Nausea.
  Participants
    Female | 7
    Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Region in which study participants have been recruited.
  participants
    Canada | 14

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Maraviroc and Rifabutin AUC 0-12/24
Description: Maraviroc pharmacokinetics: Maraviroc only AUC (h*μg/L), Maraviroc + Rifabutin AUC (h*μg/L), Rifabutin AUC (h*μg/L), 25-O-desacetyl rifabutin AUC (h*μg/L).
Time Frame: Maraviroc: 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10 and 12 hour. Rifabutin: 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hour..
Measure: Geometric Mean (90% Confidence Interval); unit: h*μg/L
Arm/Group | Maraviroc
Number analyzed (Participants) | 14
h*μg/L
  Maraviroc only AUC (h*μg/L) | 1026.2 [923.58 to 1128.82]
  Maraviroc + Rifabutin AUC (h*μg/L) | 847.0 [762.3 to 931.7]
  Rifabutin AUC (h*μg/L) | 4221.9 [3799.71 to 4644.09]
  25-O-desacetyl rifabutin AUC (h*μg/L) | 331.9 [298.71 to 365.09]

2. Primary Outcome: Maraviroc and Rifabutin C12/C24/Cmax PK Concentrations in Plasma.
Description: Maraviroc + Rifabutin pharmacokinetics: Maraviroc only Cmax (μg/L), Maraviroc only C12 (μg/L), Maraviroc + Rifabutin Cmax (μg/L), Maraviroc + Rifabutin C12 (μg/L), Rifabutin Cmax (μg/L), Rifabutin C24 (μg/L), 25-O-desacetyl rifabutin Cmax (μg/L), 25-O-desacetyl rifabutin C24 (μg/L).
Time Frame: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: μg/L
Arm/Group | Maraviroc
Number analyzed (Participants) | 14
μg/L
  Maraviroc only Cmax (μg/L) | 304.6 [274.14 to 335.06]
  Maraviroc only C12 (μg/L) | 23.3 [20.97 to 25.63]
  Maraviroc + Rifabutin Cmax (μg/L) | 239.8 [215.82 to 263.78]
  Maraviroc + Rifabutin C12 (μg/L) | 16.3 [14.67 to 17.93]
  Rifabutin Cmax (μg/L) | 542.2 [487.98 to 596.42]
  Rifabutin C24 (μg/L) | 71.2 [64.08 to 78.32]
  25-O-desacetyl rifabutin Cmax (μg/L) | 42.3 [38.07 to 46.53]
  25-O-desacetyl rifabutin C24 (μg/L) | 5.5 [4.95 to 6.05]

3. Secondary Outcome: Safety/Tolerability of the Treatments
Description: description and frequency of adverse events for all participants during the study.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 14
Participants
  Maraviroc: Number of Participants with Adverse Events | 6
  Maraviroc: Number of Participants without Adverse Events | 8
  Maraviroc + Rifabutin: Number of Participants with Adverse Events | 7
  Maraviroc + Rifabutin: Number of Participants without Adverse Events | 7

ADVERSE EVENTS:
Time Frame: 30 days.
Arm/Group | Maraviroc
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 11/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=14)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 — Pain in the areas surrounding and in the joints.
Fever (General disorders) | 2 — Increase in body temperature above normal threshold.
Headache (Nervous system disorders) | 6 — Pain occurring in the head.
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 — Pain in the participants limb muscles, occasionally in the Torso.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No